CLINICAL TRIAL: NCT03531372
Title: Efficacy and Safety of Mipolixin® Compared to Poliprotect ® in the Relief of Symptoms of Moderate Functional Dyspepsia and Heartburn: A Randomized, Double-blind, Parallel Group,Non-inferiority Clinical Study
Brief Title: Mipolixin® Compared to Poliprotect® in Moderate Functional Dyspepsia and Heartburn.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aboca Spa Societa' Agricola (Industry)
Collaborators: La Sociedad Española de Médicos de Atención Primaria (Other); Dynamic (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ABO-NB-SEM-17
Record Dates: First submitted 2018-05-09; First posted 2018-05-21 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Dyspepsia; Heartburn
MeSH Terms: conditions — Dyspepsia; Heartburn

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mipolixin® (Experimental): Mipolixin® (Advanced Natural Antacid - AdNA)
  Interventions: Device: Mipolixin®
- Poliprotect® (Active Comparator): Poliprotect® (Neobianacid)
  Interventions: Device: Poliprotect®

INTERVENTIONS:
Device: Mipolixin® — 1.55g chewable tablet 5 times a day for 2 weeks
  Other Names: Advanced Natural Antacid
  Arms: Mipolixin®
Device: Poliprotect® — 1.55 g chewable tablet 5 times a day for 2 weeks
  Other Names: Neobianacid
  Arms: Poliprotect®

SUMMARY:
Evaluation of the clinical efficacy of two medical devices, Mipolixin® and Poliprotect®, in improving the overall symptom severity of functional dyspesia and/or heartburn

ELIGIBILITY:
Inclusion Criteria:

* Ability to provide informed consent, preferably in writing or, failing that, orally in front of a witness, before any study procedure is performed.
* Male and female patients aged 18 to 75 years old (inclusive).
* Patients with symptoms of functional dyspepsia (according to the Rome IV criteria) of moderate severity (VAS score between 30 mm and 70 mm) and/or bothersome heartburn within 2 and 14 days prior to the screening/baseline visit.

  o According to the current Rome IV diagnostic criteria, functional dyspepsia is defined as one or more of the following symptoms: postprandial fullness (classified as postprandial distress syndrome), early satiation (inability to finish a normal sized meal, also classified as postprandial distress syndrome), and epigastric pain or burning (classified as epigastric pain syndrome).
* Ability of the patients (according to the investigator's opinion) to comprehend the full nature and purpose of the study including possible risks and side effects.
* Patients who agree not to alter their diet in any way for the duration of the trial and to maintain it at steady state.
* Patients who agree not to make any major lifestyle changes during the trial.
* Willingness to comply with all the study procedures and schedule.
* Chronic therapies (if not related to the gastroenterological pathologies object of the study, according to the opinion of the investigator) are allowed, if the regimen is maintained stable during the whole study.

Exclusion Criteria:

* Declines or unable to provide informed consent.

  - Disease or health condition
* Patient presenting at least one of the following symptoms or conditions at screening: anemia, chronic gastrointestinal bleeding, progressive unintentional weight loss, epigastric mass, anorexia, persistent or recurrent vomiting, dysphagia or odynophagia, porphyria, hypophosphatemia, and/or cachexia.
* Patients presenting with at least of the following gastrointestinal conditions at screening: erosive GERD, Barrett's oesophagus or oesophageal stricture, active or healing gastroduodenal ulcer (except scars), history of gastric, duodenal or esophageal surgery, symptomatic gallstone, and/or other gastrointestinal disease such as gastroenteritis, inflammatory bowel disease, celiac disease and/or colorectal cancer.
* Patients with known malignancy disease, infectious disease or severe heart or pulmonary disease.
* Patients with known severe liver or kidney disease (AST/SGOT, ALT/SGPT >2 upper limits of normal, serum creatinine >1.5 mg/dl).
* Patients with mental or metabolic disorders and any other disease that according to the physician can compromise the patient´s safety and/or patient´s study compliance.

  - Treatments
* Patients receiving any treatment (pharmacological or medical device) for heartburn or dyspeptic symptoms within the last 14 days prior to randomization.
* Patients receiving any drugs that could affect symptoms or study evaluation such antacids, PPIs, H2RAs, prokinetics, and/or gastric mucosal protectants at baseline and/or taken within the last 14 days prior to randomization.
* Patients receiving any drugs that could affect symptoms or the study as antibiotics, NSAIDs, anticholinergics and/or cholinergic agents.

Note: Patients will be asked to avoid any drugs of the above mentioned since the beginning of the study (baseline visit) until the end of the study.

* Patients under triple therapy or eradication therapy against Helicobacter pylori.
* Patients planned for long-term new therapies with anti-anxiety agents, glucocorticosteroids and anti-inflammatory agents during study period.
* Known hypersensitive or intolerance to any components of the study medical devices.
* Previous intake of any of the study medical devices.

  - Other general conditions
* Patients who are unable to understand or are unwilling to sign an informed consent form.
* Unable or unwilling to complete all required screening and/or follow-up assessments.
* Unable to understand and complete self-administered scales/questionnaires planned to be used in the study.
* Participation in interventional research studies of investigational medicinal or device products (ongoing or terminated less than 30 days before screening)
* Patients with active alcohol or drug addiction or any other condition that, in the investigator's opinion, would interfere with their ability to comply with the study requirements.
* Patients with any concurrent condition that, in the investigator's opinion, would jeopardize the safety of the patient or compliance with the protocol.
* Pregnant or nursing (lactating) women;
* Women of childbearing potential and sexually active: they must be willing to use at least one acceptable effective contraceptive measure (- progestogen-only oral hormonal contraception, where inhibition of ovulation is not the primary mode of action , - male or female condom with or without spermicide, - cap, diaphragm or sponge with spermicide). Pregnancy test will be performed at screening and at the final/premature withdrawal visit. The use of contraception in male patients is not required.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 158 (Actual)
Dates: Start 2018-04-24 (Actual); Primary Completion 2021-04-30 (Actual); Study Completion 2021-04-30 (Actual)

PRIMARY OUTCOMES:
Change in overall symptom severity from baseline (day 0) to day 14 between the two study arms | Day 0 and Day 14
  The primary endpoint is the change in the score of a visual analog scale (VAS) (from "no symptoms" to "overwhelming symptoms") used for evaluating overall symptom severity from baseline (day 0) to day 14 after treatment initiation, between the two study arms. A decrease in VAS score of at least 30% is considered as a clinically meaningful improvement, and therefore subjects achieving a decrease ≥30% in this scale will be considered as responders. The non-inferiority is considered demonstrated if the 95% confidence interval of the difference in the percentage of responders between both study arms lies within the non-inferior margin value defined of 20%.

SECONDARY OUTCOMES:
Responders from baseline to day 3 and day 7 | Day 0, Day 3 and Day 7
  Percentage of responder patients (VAS score decrease of at least 30%) on the basis of the mean change in the overall symptom severity assessed by the VAS score from baseline to day 3 and day 7 in both study arms
Self-assessment severity of individual specific symtoms | Day 0, Day 1, Day 3, Day 7 and Day 14
  Comparison between Mipolixin® and Poliprotect® in the mean change of the score of the self-assessed severity of individual specific symtoms (bothersome postprandial fullness, bothersome early satiation, bothersome epigastric pain, bothersome epigastric burning, and bothersome heartburn) rated on a 100 mm VAS (from "no symptoms" to "overwhelming symptoms") from baseline to 1 3, 7 and 14 days after treatment initiation.
Change in the score of GOS scale from baseline to day 1 | Day 0 and Day 14
  Change in the score of GOS ( Global Overall Symptom) scale from baseline to day 14 in both study arms. A decrease in GOS score ≥2 is considered as a clinically meaningful improvement, and therefore subjects achieving a decrease in overall severity score ≥2 from baseline in this scale will be considered as responders.
Incidence of AEs during study treatment | Day 0 to Day 14
  Incidence and type of adverse events (AEs) and serious adverse events (SAEs) reported during study treatment.
Incidence of AEs and clinical findings during study period | Day 0 to Day 28
  Safety will be assessed on the basis of all AEs experienced during study treatment and all observed and volunteered AEs and abnormal findings on physical examination, including vital signs throughout the study.
Patient satisfaction (treatment administration) | Day 3, Day 7 and Day 14
  Patient level of satisfaction in terms of treatment administration/posology will be assessed by means of specific questions about patient level of satisfaction after the 2-week treatment period. The response will be scored on a 4-point Likert scale from 0 to 4, as follows: 1 = "very satisfied", 2 = "quite satisfied", 3 = "somewhat satisfied", 4 = "not satisfied".
Patient satisfaction (taste) | Day 3, Day 7 and Day 14
  Patient level of satisfaction in terms of chewable tablets taste will be assessed by means of specific questions about patient level of satisfaction after the 2-week treatment period. The response will be scored on a 4-point Likert scale from 0 to 4, as follows: 1 = "very satisfied", 2 = "quite satisfied", 3 = "somewhat satisfied", 4 = "not satisfied".
Treatment compliance | Day 0 to Day 14
  Treatment compliance will be evaluated by performing the IP accountability. This data will be corroborated with the information recorded in the patient diary concerning the daily administered and missed doses.

CONTACTS AND LOCATIONS:
Locations (11):
- Spain (11):
  - CS Albuñol, Albuñol
  - CS Disset de Setembre, el Prat de Llobregat
  - CS Montesa, Madrid
  - CS Goya, Madrid
  - Primary Care Centre Eloy Gonzalo, Madrid
  - CS Comillas, Madrid
  - CS Baviera, Madrid
  - CS Las Americas, Parla
  - CS San Blas, Parla
  - CS Isabel II, Parla
  - Consultorio Local Perales de Tajuña, Perales de Tajuña